CLINICAL TRIAL: NCT01073163
Title: A Study to Assess the Effect of Treatment With Bendamustine in Combination With Rituximab on QT Interval in Patients With Advanced Indolent Non-Hodgkin's Lymphoma (NHL) or Mantle Cell Lymphoma (MCL)
Brief Title: Study to Assess the Effect of Treatment With Bendamustine in Combination With Rituximab on QT Interval in Patients With Advanced Indolent Non-Hodgkin's Lymphoma (NHL) or Mantle Cell Lymphoma (MCL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C18083/3070
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Non-Hodgkin's Lymphoma; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; Rituximab

ARMS (1):
- Bendamustine with Rituximab (Experimental): Participants were administered bendamustine intravenous (IV) infusion at 90 mg/m^2 on Days 1 and 2 of each 28-day cycle, and rituximab IV infusion at 375 mg/m^2 on Day 1 of each 28-day cycle.
  Interventions: Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Bendamustine at 90 mg/m^2 IV on Days 1 and 2 of a 28-day cycle.
  Other Names: Treakisym; Ribomustin; Levact; Treanda; SDX-105
Drug: Rituximab — Rituximab at 375 mg/m^2 IV on Day 1 of a 28-day cycle.
  Other Names: Rituxan; MabThera; IDEC-C2B8

SUMMARY:
The primary objective of this study is to assess the effect of treatment with bendamustine on cardiac repolarization as reflected by the rate-corrected QT interval by the Fridericia method (QTcF).

DETAILED DESCRIPTION:
This study was originally conducted as a substudy in a subset of patients enrolled in the phase 3 study C18083/3064/NL/MN (NCT00877006) who were randomly assigned to treatment with bendamustine in combination with rituximab (BR) and who satisfied additional eligibility criteria related to cardiac function. The objective of the substudy was to obtain results to assess the effect of bendamustine treatment on cardiac polarization and any potential changes in the QT interval (corrected by the Fridericia method [QTcF]). After a period of time, the substudy was amended to be a separate stand-alone study to ensure that an adequate number of patients were included. Patients were treated for 6, and up to 8, cycles in the stand-alone study, and efficacy and safety were also assessed. In addition, a requirement to assess the pharmacokinetics of bendamustine and rituximab when used as combination therapy was added to the objectives, to determine the potential for drug interaction between bendamustine and rituximab.

ELIGIBILITY:
Key Inclusion Criteria:

* Histopathologic confirmation of one of the following CD20+ B-cell non-Hodgkin's lymphomas. Tissue diagnostic procedures must be performed within 6 months of study entry and with biopsy material available for review:

  * follicular lymphoma (grade 1 or 2)
  * immunoplasmacytoma/immunocytoma (Waldenstrom's macroglobulinemia)
  * splenic marginal zone B-cell lymphoma
  * extra-nodal marginal zone lymphoma of mucosa associated lymphoid tumor (MALT) type
  * nodal marginal zone B-cell lymphoma
  * mantle cell lymphoma
* Meets one of the following need-for-treatment criteria (with the exception of mantle cell lymphoma for which treatment is indicated):

  * presence of at least one of the following B-symptoms:

    1. fever (>38ºC) of unclear etiology
    2. night sweats
    3. weight loss of greater than 10% within the prior 6 months
  * large tumor mass (bulky disease)
  * presence of lymphoma-related complications, including narrowing of ureters or bile ducts, tumor-related compression of a vital organ, lymphoma induced pain, cytopenias related to lymphoma/leukemia, splenomegaly, pleural effusions, or ascites
  * hyperviscosity syndrome due to monoclonal gammopathy
* CD20-positive B cells in lymph node biopsy or other lymphoma pathology specimen
* No prior treatment. Patients on "watch and wait" may enter the study if a recent biopsy (obtained within the last 6 months) is available.
* Adequate hematologic function (unless abnormalities related to lymphoma infiltration of the bone marrow or hypersplenism due to lymphoma) as follows:

  * hemoglobin of >= 10.0 g/dL
  * absolute neutrophil count (ANC) >=1.5*10^9/L
  * platelet count >=100*10^9/L
* Bidimensionally measurable disease (field not previously radiated)
* Able to provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status <=2
* Estimated life expectancy >=6 months
* Serum creatinine of <=2.0 mg/dL or creatinine clearance >=50 mL/min
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5* upper limit of normal (ULN), and alkaline phosphatase and total bilirubin within normal limits
* Left ventricular ejection fraction (LVEF) >=50% by multiple gated acquisition scan (MUGA) or cardiac echocardiogram (ECHO), prior for any patient to be treated with rituximab/cyclophosphamide/doxorubicin/vincristine/prednisolone (R-CHOP)
* A medically accepted method of contraception to be used by women of childbearing potential (not surgically sterile or at least 12 months naturally postmenopausal)
* Men capable of producing offspring and not surgically sterile must practice abstinence or use a barrier method of birth control

Key Exclusion Criteria:

* Chronic lymphocytic leukemia, small lymphocytic lymphoma (SLL), or grade 3 follicular lymphoma
* Transformed disease. Bone marrow blasts are permitted, however, transformed disease indicating leukemic involvement is not permitted
* Central nervous system (CNS) lymphomatous involvement or leptomeningeal lymphoma
* Prior radiation for non-Hodgkin's lymphoma (NHL), except for a single course of locally delimited radiation therapy with a radiation field not exceeding 2 adjacent lymph node regions
* Active malignancy, other than NHL, within the past 3 years except for localized prostate cancer treated with hormone therapy, cervical carcinoma in situ, breast cancer in situ, or non-melanoma skin cancer following definitive treatment
* New York Heart Association (NYHA) Class III or IV heart failure, arrhythmias or unstable angina, electrocardiographic evidence of active ischemia or active conduction system abnormalities, or myocardial infarction within the last 6 months. (Prior to study entry, ECG abnormalities at screening must be documented by the investigator as not medically relevant)
* Known human immunodeficiency virus (HIV) positivity
* Active hepatitis B or hepatitis C infection (Hepatitis B surface antigen testing required)
* Women who are pregnant or lactating
* Corticosteroids for treatment of lymphoma within 28 days of study entry. Chronically administered low-dose corticosteroids (e.g., prednisone ≤20 mg/day) for indications other than lymphoma or lymphoma-related complications are permitted
* Any serious uncontrolled, medical or psychological disorder that would impair the ability of the patient to receive therapy
* Any condition which places the patient at unacceptable risk or confounds the ability of the investigators to interpret study data
* Any other investigational agent within 28 days of study entry
* Known hypersensitivity to bendamustine, mannitol, or other study-related drugs
* The patient has Ann Arbor stage I disease
* The patient has a history of congenital long QT syndrome
* The patient has a history of cardiac disease with significant potential for QT prolongation
* The patient has screening electrocardiography (ECG) on Day 1 of Cycle 1 with QTcF interval >450 ms that is confirmed by a second ECG. If the QTcF interval is >450 ms on both ECGs, the ECGs will be sent to eResearch Technology, Inc. (ERT), the Central ECG Reader vendor, for an overread (with 24-hour turn around time) and ERT will make a final decision on enrollment
* The patient has serum potassium or magnesium less than the lower limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (43):
- United States (36):
  - Hematology Oncology Physicans Extenders Group, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - St. Jude Heritage Medical Group, Fullerton, California
  - Comprehensive Cancer Center, Palm Springs, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Memorial Cancer Institute, Hollywood, Florida
  - Cancer Centers of Florida, Orlando, Florida
  - MD Anderson Cancer Cnt Orlando, Orlando, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - St Francis Cancer Research Foundation, Beech Grove, Indiana
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - LSU Health Sciences Center - Shreveport, Shreveport, Louisiana
  - MaineGeneral Medical Center, Augusta, Maine
  - Missouri Cancer Associates, Columbia, Missouri
  - Kansas City Cancer Center, Kansas City, Missouri
  - UNM Cancer Center/New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Interlakes Foundation, Inc, Rochester, New York
  - SUNY Upstate / Upstate Medical University, Syracuse, New York
  - Willamette Valley Cancer Center, Springfield, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Inc., Philadelphia, Pennsylvania
  - Charleston Hematology Oncology, PA, Charleston, South Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Oncology, P.A., Fort Worth, Texas
  - Cancer Care Center of South Texas, San Antonio, Texas
  - Texas Oncology, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Cancer Outreach Asscociates, PC, Richlands, Virginia
  - Cancer Care Northwest-South, Spokane, Washington
  - Northwest Cancer Specialists, PC, Vancouver, Washington
  - West Virginia University School of Medicine, Morgantown, West Virginia
- Australia (5):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Alfred Hospital, Melbourne, Victoria
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Ottawa Hospital - General Campus, Ottawa, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-five patients were screened for this study; 8 did not meet eligibility criteria, and 3 were not enrolled for other reasons.
Period: Overall Study
Arm/Group | Bendamustine With Rituximab
Started | 54
Enrolled But Not Treated | 1
Treated With <6 Cycles | 4
Treated With >=6 Cycles | 49
Completed | 51 (Patients completed study)
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Disease Progression | 1
Not completed — Early termination | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years]
  AgeContinuous | 62.9 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 49
  Other | 4
Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Scale scores were: 0=fully active, able to carry on all pre-disease performance without restriction; 1=restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=dead.
  participants
    Score=0 | 29
    Score=1 | 20
    Score=2 | 5
    Score=3 | 0
    Score=4 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in QT Interval as Corrected by the Fridericia Method (QTcF) at End of Infusion
Description: On Day 2 of Cycle 1, three electrocardiograms (ECGs) were collected 15 minutes prior to any study drug administration. The baseline ECG interval value was obtained by averaging these 3 ECGs, and was compared to the average of the 3 ECGs taken on treatment with bendamustine at the end of the infusion.
Time Frame: Baseline ECGs (Day 2 of Cycle 1): 15 minutes prior to bendamustine infusion. Postinfusion ECGs (Day 2 of Cycle 1): at the end of the 30-minute infusion.
Population: ECG Analysis Set: all enrolled participants in study who received at least 1 dose of study drug and with at least 1 available baseline and 1 on-treatment ECG; n=number of participants with measurement at given time point.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 53
milliseconds (ms)
  Baseline, n=53 | 410.4 (23.6)
  End of Infusion, n=52 | 6.7 (10.3) [9.1 to 4.3]

2. Secondary Outcome: Mean Change From Baseline in QTcF at 1 Hour Postinfusion
Description: On Day 2 of Cycle 1, three ECGs were collected 15 minutes prior to any study drug administration. The baseline ECG interval value was obtained by averaging these 3 ECGs, and was compared to the average of the 3 ECGs taken on treatment with bendamustine 1 hour postinfusion.
Time Frame: Baseline ECGs (Day 2 of Cycle 1): 15 minutes prior to bendamustine infusion. Postinfusion ECGs (Day 2 of Cycle 1): 1 hour postinfusion.
Population: ECG Analysis Set: all enrolled participants in study who received at least 1 dose of study drug and with at least 1 available baseline and 1 on-treatment ECG.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 53
ms
  Baseline | 410.4 (23.6)
  1 Hour Postinfusion | 4.1 (9.8)

3. Secondary Outcome: Number of Participants With QTcF New Outlier Events at End of Infusion and 1 Hour Postinfusion
Description: Participants were considered to have an outlier ECG value based on the most extreme value across each of the time points. "New" means not present at baseline and becomes present on at least 1 on-treatment ECG time point. A participant had a new outlier event (500) if the maximum QTcF was >500 ms while their baseline was <=500 ms, or had an outlier event (480) if the maximum QTcF was >480 ms while their baseline was <= 480 ms. QTcF in the 30-60 ms or >60 ms categories were also considered outliers.
Time Frame: Baseline ECGs (Day 2 of Cycle 1): 15 minutes prior to bendamustine infusion. Postinfusion ECGs (Day 2 of Cycle 1): at the end of the 30-minute infusion and 1 hour postinfusion.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 53
participants
  QTcF New >500 ms at End of Infusion; n=52 | 0
  QTcF New >500 ms 1 Hour Postinfusion; n=53 | 0
  QTcF New >480 ms at End of Infusion; n=52 | 1
  QTcF New >480 ms 1 Hour Postinfusion; n=53 | 0
  QTcF New >60 ms at End of Infusion; n=52 | 0
  QTcF New >60 ms 1 Hour Postinfusion; n=53 | 0
  QTcF New 30-60 ms at End of Infusion; n=52 | 0
  QTcF New 30-60 ms 1 Hour Postinfusion; n=53 | 0

4. Secondary Outcome: Number of Participants With New Onset ECG Waveform Morphological Changes
Description: The core ECG laboratory cardiologist assessed all leads in the ECGs and defined morphological changes. Changes from baseline (looking at each of the 3 ECGs at Day 2 Cycle 1 individually and the ECGs at all on-treatment time points individually) were noted for the following events: atrial fibrillation or flutter; second degree heart block; third degree heart block; complete right bundle branch block; complete left bundle branch block; ST segment depression; T wave abnormalities (negative T waves only); myocardial infarction pattern; any new abnormal U waves.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 53
participants | 0

5. Secondary Outcome: Number of Participants With Treatment-Emergent Cardiac Disorders
Description: Number of participants with cardiac disorders overall, with severity from grades 1 (mild) to grade 4 (severe), according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 (grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening, grade 5= death). Participants may have reported more than 1 event.
Time Frame: Adverse events were collected throughout the study and up to 30 days after the last dose of study drug. The median number of 28-day cycles was 6.0. The median duration of the treatment period was 143 days.
Population: Safety Analysis Set: enrolled participants who received 1 or more doses of study drug.
Measure: Number; unit: participants
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 53
participants
  ECG QT prolonged: Overall | 3
  ECG QT prolonged: Grade >/=3 | 2
  Blood pressure decreased: Overall | 1
  Blood pressure decreased: Grade >/=3 | 1
  Cardiac murmur: Overall | 1
  Cardiac murmur: Grade >/=3 | 0
  ECG ST segment abnormal: Overall | 1
  ECG ST segment abnormal: Grade >/=3 | 0
  Heart rate irregular: Overall | 1
  Heart rate irregular: Grade >/=3 | 0
  Palpitations: Overall | 2
  Palpitations: Grade >/=3 | 0
  Arteriosclerosis coronary artery: Overall | 1
  Arteriosclerosis coronary artery: Grade >/=3 | 0
  Atrial fibrillation: Overall | 1
  Atrial fibrillation: Grade >/=3 | 0
  Cardiac failure congestive: Overall | 1
  Cardiac failure congestive: Grade >/=3 | 0
  Left ventricular dysfunction: Overall | 1
  Left ventricular dysfunction: Grade >/=3 | 1
  Sinus tachycardia: Overall | 1
  Sinus tachycardia: Grade >/=3 | 0
  Tachycardia: Overall | 1
  Tachycardia: Grade >/=3 | 0

6. Secondary Outcome: Change From Baseline in QTcF at Maximum Concentration (Cmax) of Bendamustine and Its Metabolites (M3 and M4)
Description: Results from a pharmacokinetic-pharmacodynamic model to show the relationship of the overall predicted change from Baseline in QTcF at the average Cmax of bendamustine and its metabolites M3 and M4.
Time Frame: as for outcome 3
Population: Pharmacokinetic-pharmacodynamic Analysis Set: all enrolled participants in study who received at least 1 dose of study drug and with at least 1 available baseline and 1 on-treatment ECG and at least 1 ECG with a time-matched plasma concentration pair.
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 51
ms
  Bendamustine | 5.4097 [NA to 7.5670] — One-sided confidence interval was calculated.
  Metabolite M3 | 5.9995 [NA to 8.8415] — One-sided confidence interval was calculated.
  Metabolite M4 | 7.1390 [NA to 10.0904] — One-sided confidence interval was calculated.

7. Secondary Outcome: Model-predicted Bayesian Bendamustine Clearance in the Presence of Rituximab
Description: Boxplots of model-predicted Bayesian bendamustine clearance (CL) values in the presence of rituximab were generated based on the administered bendamustine doses, rate of infusion, and sample times.
Time Frame: Day 1 of Cycle 1: prior to start of bendamustine infusion, immediately postinfusion, 15 minutes and 30 minutes postinfusion. Day 2 of Cycle 1: 15 minutes prior to start of bendamustine infusion, 15 minutes, 30 minutes, 1, 3, and 5 hours postinfusion.
Population: Pharmacokinetic Analysis Set: all enrolled participants in study who received at least 1 dose of study drug and with at least 1 quantifiable bendamustine plasma concentration.
Measure: Median (Full Range); unit: L/h
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 49
L/h | 32.9 (12.8) [0.9 to 58.5]

8. Secondary Outcome: Rituximab Concentrations at 0.5 Hours, 24 Hours, and 7 Days Postinfusion
Time Frame: Day 1 of Cycle 1: prior to start of rituximab infusion, immediately postinfusion. Day 2 of Cycle 1: 15 minutes prior to the start of the bendamustine infusion. Day 7 and Day 14: anytime. Day 1 of Cycle 2: prior to start of rituximab infusion.
Population: Pharmacokinetic Analysis Set: all enrolled participants in study who received at least 1 dose of study drug and with at least 1 quantifiable serum concentration of rituximab.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 19
mcg/mL
  0.5 Hours Postinfusion; n=19 | 173.0 [74.5 to 299.0]
  24 Hours Postinfusion; n=19 | 105.0 [4.62 to 176.0]
  7 Days Postinfusion; n=17 | 30.5 [0.256 to 73.3]

9. Secondary Outcome: Percentage of Participants With Complete Response (CR)
Description: Complete response, as defined by the International Working Group (IWG) Revised Response Criteria For Malignant Lymphoma. Results are presented for participants with non-Hodgkin lymphoma and mantle cell lymphoma as well as all participants.
Time Frame: The median number of 28-day cycles was 6.0. The median duration of the treatment period was 143 days.
Population: Full Analysis Set: all enrolled participants who received at least 1 dose of both bendamustine and rituximab and who had both a baseline and at least 1 postbaseline tumor response evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Non-Hodgkin Lymphoma: Participants with non-Hodgkin Lymphoma were administered bendamustine intravenous (IV) infusion at 90 mg/m^2 on Days 1 and 2 of each 28-day cycle, and rituximab IV infusion at 375 mg/m^2 on Day 1 of each 28-day cycle.
- Mantle Cell Lymphoma: Participants with mantle cell lymphoma were administered bendamustine intravenous (IV) infusion at 90 mg/m^2 on Days 1 and 2 of each 28-day cycle, and rituximab IV infusion at 375 mg/m^2 on Day 1 of each 28-day cycle.
- Total: All participants administered bendamustine intravenous (IV) infusion at 90 mg/m^2 on Days 1 and 2 of each 28-day cycle, and rituximab IV infusion at 375 mg/m^2 on Day 1 of each 28-day cycle.
Arm/Group | Non-Hodgkin Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 40 | 11 | 51
percentage of participants | 40 [24.9 to 56.7] | 55 [23.4 to 83.3] | 43 [29.3 to 57.8]

10. Secondary Outcome: Percentage of Participants With Overall Response
Description: Overall Response was comprised of those participants who had Complete Response (CR) plus those who had Partial Response (PR), as defined by the International Working Group (IWG) Revised Response Criteria For Malignant Lymphoma. Results are presented for participants with non-Hodgkin lymphoma and mantle cell lymphoma as well as all participants.
Time Frame: The median number of 28-day cycles was 6.0. The median duration of the treatment period was 143 days.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Hodgkin Lymphoma | Mantle Cell Lymphoma | Total
Number analyzed (Participants) | 40 | 11 | 51
percentage of participants | 93 [79.6 to 98.4] | 100 [71.5 to 100.0] | 94 [83.8 to 98.8]

11. Secondary Outcome: Overview of Adverse Events
Description: Adverse event (AE)=any untoward medical occurrence in a patient administered study drug that develops or worsens in severity during the conduct of a clinical study of a pharmaceutical product and does not necessarily have a causal relationship to the study drug. Treatment-related AEs=those that began or worsened after treatment with study drug. AE severity was graded according to the National Cancer Institute's Common Terminology Criteria for AEs (grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening, grade 5= death). Relationship of an AE to study drug was categorized as definite, probable, possible, unlikely, or not related. Serious AE (SAE)=one that occurred at any dose that resulted in any of the following outcomes or actions: death; a life-threatening adverse event; inpatient hospitalization or prolongation of existing hospitalization; a persistent or significant disability/incapacity; a congenital anomaly/birth defect; or an otherwise important medical event.
Time Frame: as for outcome 5
Population: Safety Analysis Set: enrolled participants who received 1 or more doses of study drug.
Measure: Number; unit: participants
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 53
participants
  Any adverse event | 53
  Severe adverse events (grade 3, 4, 5) | 33
  Treatment-related adverse events | 52
  Deaths | 1
  Other serious adverse events | 14
  Withdrawn from study due to adverse events | 1

12. Secondary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status at Endpoint
Description: The investigator assessed each patient's ECOG performance status according to the ECOG scale at screening, on Day 1 of each treatment cycle, and at the end-of-treatment visit. Scale scores were: 0=fully active, able to carry on all pre-disease performance without restriction; 1=restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=dead. Any change in score to a higher value signifies worsening, and any change to a lower value signifies improvement.
Time Frame: End of study. The median number of 28-day cycles was 6.0. The median duration of the treatment period was 143 days.
Population: Safety Analysis Set: enrolled participants who received 1 or more doses of study drug.
Measure: Number; unit: participants
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 53
participants
  Improved | 10
  Stayed the same | 35
  Worsened | 8

13. Secondary Outcome: Worst Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 Grades for Hematology Laboratory Tests Results Overall
Description: Grade 1=Mild, 2=Moderate, 3=Severe/medically significant, 4=Life-threatening. Overall is defined as the worst postbaseline grade value for each patient and laboratory test across all cycles. Only postbaseline grades are summarized. If absolute neutrophil count (ANC) and neutrophils absolute (ABS) were both measured, the worse grade value from the two was summarized. Otherwise the worst ANC grade value or the worst neutrophils ABS grade value was summarized. WBC=white blood cell; LLN=lower limit of normal
Time Frame: as for outcome 5
Population: Safety Analysis Set: enrolled participants who received 1 or more doses of study drug.
Measure: Number; unit: participants
Arm/Group | Bendamustine With Rituximab
Number analyzed (Participants) | 53
participants
  ANC, Grade 1: <LLN - 1.5*10^9/L | 5
  ANC, Grade 2: <1.5 - 1.0*10^9/L | 12
  ANC, Grade 3: <1.0 - 0.5*10^9/L | 11
  ANC, Grade 4: <0.5*10^9/L | 12
  ANC, Grade 1-4 | 40
  Hemoglobin, Grade 1: <LLN - 100 g/L | 36
  Hemoglobin, Grade 2: <100 - 80 g/L | 12
  Hemoglobin, Grade 3: <80 - 65 g/L | 1
  Hemoglobin, Grade 4: <65 g/L | 0
  Hemoglobin, Grade 1-4 | 49
  Lymphocytes ABS, Grade 1: <LLN - 0.8*10^9/L | 0
  Lymphocytes ABS, Grade 2: <0.8 - 0.5*10^9/L | 2
  Lymphocytes ABS, Grade 3: <0.5 - 0.2*10^9/L | 13
  Lymphocytes ABS, Grade 4: <0.2*10^9/L | 22
  Lymphocytes ABS, Grade 1-4 | 37
  Platelets, Grade 1: <LLN - 75.0*10^9/L | 19
  Platelets, Grade 2: <75.0 - 50.0*10^9/L | 9
  Platelets, Grade 3: <50.0 - 25.0*10^9/L | 3
  Platelets, Grade 4: <25.0*10^9 /L | 1
  Platelets, Grade 1-4 | 32
  WBC, Grade 1: <LLN - 3.0*10^9/L | 9
  WBC, Grade 2: <3.0 - 2.0*10^9/L | 19
  WBC, Grade 3: <2.0 - 1.0*10^9/L | 15
  WBC, Grade 4: <1.0*10^9/L | 5
  WBC, Grade 1-4 | 48

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study and up to 30 days after the last dose of study drug. The median number of 28-day cycles was 6.0. The median duration of the treatment period was 143 days.
Description: Safety Analysis Set: enrolled participants who received 1 or more doses of study drug.
Arm/Group | Bendamustine With Rituximab
Serious Adverse Events (participants affected / at risk) | 14/53
Other Adverse Events (participants affected / at risk) | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine With Rituximab (N=53)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Appendix disorder (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chills (General disorders) | 1 (2)
Pyrexia (General disorders) | 2 (3)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine With Rituximab (N=53)
Anaemia (Blood and lymphatic system disorders) | 6 (18)
Neutropenia (Blood and lymphatic system disorders) | 19 (50)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (18)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 5 (9)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 22 (28)
Diarrhoea (Gastrointestinal disorders) | 16 (21)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5)
Mouth ulceration (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 38 (56)
Stomatitis (Gastrointestinal disorders) | 7 (8)
Vomiting (Gastrointestinal disorders) | 16 (21)
Asthenia (General disorders) | 3 (3)
Chills (General disorders) | 7 (9)
Fatigue (General disorders) | 27 (38)
Feeling cold (General disorders) | 3 (3)
Influenza like illness (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 4 (6)
Pain (General disorders) | 6 (6)
Pyrexia (General disorders) | 12 (20)
Drug hypersensitivity (Immune system disorders) | 8 (10)
Nasopharyngitis (Infections and infestations) | 4 (4)
Oral herpes (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (9)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 19 (46)
Electrocardiogram QT prolonged (Investigations) | 3 (4)
Weight decreased (Investigations) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Dizziness (Nervous system disorders) | 5 (6)
Dysgeusia (Nervous system disorders) | 9 (10)
Headache (Nervous system disorders) | 9 (10)
Anxiety (Psychiatric disorders) | 5 (6)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 12 (13)
Nocturia (Renal and urinary disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 7 (9)
Hot flush (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator/Institution must submit proposed publication to Sponsor for review within a prespecified number of days before submission for publication. If Sponsor's review shows that potentially patentable subject matter would be disclosed, publication/public disclosure shall be delayed to enable Sponsor, or Sponsor's designees, to file necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.